CLINICAL TRIAL: NCT00574132
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Efficacy and Safety Trial of Bapineuzumab (AAB-001, ELN115727) In Patients With Mild to Moderate Alzheimer's Disease Who Are Apolipoprotein E4 Non- Carriers.
Brief Title: Bapineuzumab in Patients With Mild to Moderate Alzheimer's Disease (ApoE4 Non-Carrier)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JANSSEN Alzheimer Immunotherapy Research & Development, LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELN115727-301
Record Dates: First submitted 2007-12-10; First posted 2007-12-17 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — bapineuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Bapineuzumab 0.5 mg/kg (Experimental): infusion every 13 weeks for a total of 6 infusions
  Interventions: Drug: Bapineuzumab 0.5 mg/kg
- Placebo Control (Placebo Comparator): infusion every 13 weeks for a total of 6 infusions.
  Interventions: Drug: Placebo Control
- Bapineuzumab 1.0 m/kg (Experimental): infusion every 13 weeks for a total of 6 infusions.
  Interventions: Drug: Bapineuzumab 1.0 m/kg

INTERVENTIONS:
Drug: Bapineuzumab 0.5 mg/kg — infusion every 13 weeks for a total of 6 infusions
  Other Names: AAB-001
  Arms: Bapineuzumab 0.5 mg/kg
Drug: Placebo Control — given by infusion every 13 weeks for a total of 6 infusions.
  Arms: Placebo Control
Drug: Bapineuzumab 1.0 m/kg — infusion every 13 weeks for a total of 6 infusions
  Other Names: AAB-001
  Arms: Bapineuzumab 1.0 m/kg

SUMMARY:
This is a multicenter, double-blind, placebo controlled, randomized, outpatient multiple dose study in male and female patients ages 50 to less than 89 years with mild to moderate AD. Approximately 230 study sites in the US and Canada and up to 35 sites outside of North America will be involved. Patients will be randomized to receive either bapineuzumab or placebo. Each patient's participation will last approximately 1.5 years.

Bapineuzumab is a humanized monoclonal antibody, which binds to and clears beta amyloid peptide, and is designed to provide antibodies to beta amyloid directly to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD
* Age from 50 to less than 89
* Mini-Mental Status Exam score of 16-26 inclusive
* Brain magnetic resonance imaging (MRI) scan consistent with the diagnosis of AD
* Stable doses of medications (cholinesterase inhibitors and memantine allowed)
* Caregiver able to attend all clinic visits with patient

Exclusion Criteria:

* Significant neurological disease other than AD
* Major psychiatric disorder
* Significant systemic illness
* History of stroke or seizure, autoimmune disease, myocardial infarction within the last 2 years
* Smoking greater than 20 cigarettes per day
* Anticonvulsants, anti-Parkinson's, anticoagulant, or narcotic medications
* Prior treatment experimental immunotherapeutics or vaccines for AD
* Women of childbearing potential
* Presence of pacemakers, CSF shunts, or foreign metal objects in the eyes, skin or body

Ages: 50 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1331 (Actual)
Dates: Start 2007-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Cognitive and Functional | 18 months

SECONDARY OUTCOMES:
Cognitive and Global | 18 months
Imaging and biochemical biomarkers of disease status | 18 months

CONTACTS AND LOCATIONS:
Locations (251):
- United States (219):
  - University of Alabama Hospital (UAB), Birmingham, Alabama
  - Dedicated Clinical Research, Inc., Goodyear, Arizona
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - HOPE Research Institute, LLC, Phoenix, Arizona
  - Banner Research Institute, Sun City, Arizona
  - University of Arizona College of Medicine, Health Science Center, Tucson, Arizona
  - Northwest Neurospecialists, PLLC, Tucson, Arizona
  - Clinical Trials Inc., Little Rock, Arkansas
  - East Bay Physicians Medical Group, Berkeley, California
  - AVI Clinical Research, Carson, California
  - ATP Clinical Research, Inc, Costa Mesa, California
  - Pharmacology Research Institute, Encino, California
  - Margolin Brain Institute, Fresno, California
  - Neurology Center of North Orange County, Fullerton, California
  - Integrated Medical and Behavioral Associates, Glendale, California
  - Sun Valley Behavioral Medical Center, Imperial, California
  - Coordinated Clinical Research, La Jolla, California
  - University of California San Diego/Shela Marcos Alzheimer's Disease Research Center, La Jolla, California
  - Senior Clinical Trials, Laguna Hills, California
  - Collaborative Neuroscience Network, Long Beach, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Vintage Institute for Clinical Research, Inc, Los Angeles, California
  - UCLA Department of Neurology, Los Angeles, California
  - Synergy Research, National City, California
  - Pharmacology Research Institute, Newport Beach, California
  - The Neurology Center, Oceanside, California
  - University of California, Irvine Medical Center, Orange, California
  - Neuro-Therapeutics Inc., Pasadena, California
  - The Southwest Institute for Clinical Research, Inc., Rancho Mirage, California
  - Sutter Neuroscience Medical Group, Sacramento, California
  - University of California, Davis, Alzheimer's Disease Center, Sacramento, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Neurological Research Institute, Santa Monica, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Diablo Clinical Research, Inc, Walnut Creek, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Mile High Research Center, Denver, Colorado
  - Advanced Neurosciences Research, LLC, Fort Collins, Colorado
  - Associated Neurologists, PC, Danbury, Connecticut
  - Associated Neurologists of Southern CT, P.C., Fairfield, Connecticut
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Yale University School of Medicine, Alzheimer's Disease Research Unit, New Haven, Connecticut
  - Research Center for Clinical Studies, Inc, Norwalk, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - JEM Research, LLC, Atlantis, Florida
  - Bradenton Research Center, Inc, Bradenton, Florida
  - Quantum Laboratories, Inc., Deerfield Beach, Florida
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Neurologic Consultants, P.A., Fort Lauderdale, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Clinical Physiology Associates, Inc., Fort Myers, Florida
  - Emerald Coast Mood & Memory, PA., Fort Walton Beach, Florida
  - MD Clinical, Hallandale, Florida
  - Sunrise Clinical Research, Inc., Hollywood, Florida
  - Mayo Clinic College of Medicine, Jacksonville, Florida
  - Neurology Associates, Maitland, Florida
  - Melbourne International Medicine Associates, MIMA, Melbourne, Florida
  - Pharmax Research Clinic, LLC, Miami, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Allied Clinical Trials, Inc., Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Compass Research, LLC, Orlando, Florida
  - Palm Beach Neurological Center/Advanced Research Consultants, Palm Beach Gardens, Florida
  - Broward Research Group, Inc., Pembroke Pines, Florida
  - Neurostudies, Inc, Port Charlotte, Florida
  - Roskamp Institute, Sarasota, Florida
  - Miami Research Associates, South Miami, Florida
  - Meridien Research, St. Petersburg, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Johnnie B. Byrd Sr. Alzheimer's Center and Research Institute, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - University of South Florida Suncoast Alzheimer's and Gerontology Center, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Emory University/School of Medicine, Atlanta, Georgia
  - MS Center of Atlanta, Atlanta, Georgia
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Medical Research and Health Education Foundation, Inc., Columbus, Georgia
  - Dekalb Neurology Associates, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Alexian Brothers Neurosciences Institute, Elk Grove Village, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Southern Illinois University, School of Medicine, Springfield, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Kansas Multi-Specialist Group, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mid America Neuroscience Institute, Lenexa, Kansas
  - Associates in Neurology, PSC, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - Louisana State University Health Sciences Center, Shreveport, Louisiana
  - J. Gary Booker, MD, APMC, Shreveport, Louisiana
  - Maine Medical Partners Neurology, Scarborough, Maine
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - CBH Health, LLC, Rockville, Maryland
  - McLean Hospital, Belmont, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - ActivMed Practices and Research, Inc, Haverhill, Massachusetts
  - Neurocare, Inc., Newton, Massachusetts
  - Neuroscience Research of the Berkshires, Pittsfield, Massachusetts
  - Donald S. Marks, MD, P.C., Plymouth, Massachusetts
  - Memory Wellness Clinic, Springfield, Massachusetts
  - Springfield Neurology Associates, Springfield, Massachusetts
  - Coastal Research Associates, Inc., Weymouth, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Saint Mary's Health Care, Grand Rapids, Michigan
  - Borgess Medical Center/Borgess Research Institute, Kalamazoo, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Precise Research Centers, Flowood, Mississippi
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Saint Luke's Hospital, Mid America Brain and Stroke Institute, Kansas City, Missouri
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - St. Louis University School of Medicine, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Deaconess Billings Clinical Research Center, Billings, Montana
  - Advanced Neurology Specialists, Great Falls, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Coastal Neurology, PA, Dover, New Hampshire
  - Dartmouth Hitchcock Medical Center, Dept of Neurology, Lebanon, New Hampshire
  - Comprehensive Clinical Research, Berlin, New Jersey
  - The Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - The NeuroCognitive Institute, Mount Arlington, New Jersey
  - Alzheimer's Research Corporation (ARC), Paterson, New Jersey
  - Princeton Medical Institute, Princeton, New Jersey
  - University of Medicine and Dentistry of New Jersey, Stratford, New Jersey
  - Shore Neurology, P.A., Toms River, New Jersey
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - University of New Mexico, Health Sciences Center, Albuquerque, New Mexico
  - Upstate Clinical Research, LLC, Albany, New York
  - Neurological Associates of Albany, P.C., Albany, New York
  - Neuroscience Research Center at Albany Medical Center, Albany, New York
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Five Towns Neuroscience Research, Cedarhurst, New York
  - Advanced Bio-Behavioral Sciences, Elmsford, New York
  - Empire Neurology, PC, Latham, New York
  - Neurological Care of CNY, Liverpool, New York
  - Parker Jewish Institute for Health Care & Rehabilitation, New Hyde Park, New York
  - NYU School of Medicine/Psychiatry, New York, New York
  - Mt. Sinai School of Medicine, New York, New York
  - Columbia University/Medical Center, New York, New York
  - Dent Neurologic Institute, New York, New York
  - Nathan S. Kline Institute for Psychiatric Research, Orangeburg, New York
  - University of Rochester Medical Center @ Monroe Community Hospital, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Clinical Trials of America, Inc, Hickory, North Carolina
  - New Hope Clinical Research, Hickory, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Rakesh Ranjan, M.D. & Associates, Inc., Beachwood, Ohio
  - Neuro-Behavioral Clinical Research, Inc, Canton, Ohio
  - NeuroCare Center, Inc, Canton, Ohio
  - University Memory and Aging Center University Hospitals of Cleveland/Case Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Neurology Specialists, Inc., Dayton, Ohio
  - Neurology and Neuroscience Center of Ohio, Toledo, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Red River Medical Research Center, LLC, Oklahoma City, Oklahoma
  - Providence Medical Group-Medford Neurology, Medford, Oregon
  - Summit Research Group, Inc., Portland, Oregon
  - Providence Health Service System, AD Center, Brain Institute, Portland, Oregon
  - Oregon Health & Sciences University, Portland, Oregon
  - Abington Neurological Associates, Ltd, Abington, Pennsylvania
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Penn Memory Center, Philadelphia, Pennsylvania
  - Jefferson Hospital for Neuroscience, Philadelphia, Pennsylvania
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Mood and Memory Research Institute, East Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Medical University of South Carolina, North Charleston, South Carolina
  - Avera Research Institute, Sioux Falls, South Dakota
  - Neurology Clinic, PC, Cordova, Tennessee
  - Psychiatric Consultants, PC, Franklin, Tennessee
  - East Tennessee State University, Johnson City, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Senior Adults Specialty Research (SASR), Austin, Texas
  - Texas Neurology, PA, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - University of North Texas/Health Sciences Center-Fort Worth, Fort Worth, Texas
  - Claghorn-Lesem Research Clinic, Ltd., Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - Integra Clinical Research, LLC, San Antonio, Texas
  - Grayline Clinical Drug Trials, Inc, Wichita Falls, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - University of Utah, Dept of Neurology, Salt Lake City, Utah
  - The Memory Clinic, Bennington, Vermont
  - Fletcher Allen Health Care, Burlington, Vermont
  - Innovative Clinical Research Center, Alexandria, Virginia
  - University of Virginia, Charlottesville, Virginia
  - Alliance Research Group, LLC, Richmond, Virginia
  - University of Washington Veterans Affairs, Seattle, Washington
  - Pacific Medical Centers, Seattle, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - University of Wisconson Medical School of Medicine and Public Health, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Independent Pyschiatric Consultants, Waukesha, Wisconsin
- Austria (2):
  - Medizinische Universität Graz, Graz, Styria
  - Medizinische Universität Wien, Vienna, Vienna
- Canada (18):
  - University of Calgary, Foothills Medical Centre, Calgary, Alberta
  - Medical Arts Health Research Group, Kamloops, British Columbia
  - Medical Arts Health Research Group, Kelowna, British Columbia
  - Medical Arts Health Research Group, Penticton, British Columbia
  - University of British Columbia (UBC) Hospital, Vancouver, British Columbia
  - Hotel Dieu Hospital/Queens University Memorial Clinics, Kingston, Ontario
  - Saint Joseph's Health Care London, Saint Joseph's Hospital, London, Ontario
  - Parkwood Hospital, London, Ontario
  - Bruyere Continuing Care, Ottawa, Ontario
  - Kawartha Regional Memory Clinic, Peterborough, Ontario
  - Neurology Research Inch./Toronto Memory Program, Toronto, Ontario
  - Toronto Centre for Memory and Aging, Toronto, Ontario
  - Ontario Shores Centre for Mental Health Scienes, Whitby, Ontario
  - Neuro Rive-Sud Memory Clinic, Greenfield Park, Quebec
  - Hopital Maisonneuve-Rosemont, Comite d' ethique de la recherche, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
  - Douglas Mental Health University Institute, Verdun, Quebec
- Germany (12):
  - Universitätsklinik Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinik Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinik Ulm, Ulm, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Günzburg, Bavaria
  - Ludwig-Maximilians-Universität München, München, Bavaria
  - Klinikum Rechts der Isar der Technischen Universität München, München, Bavaria
  - Universitätsklinikum Regensburg, Regensburg, Byern
  - UKE Hamburg, Hamburg, Hamburg
  - Saint Josefs Hospital, Bochum, North Rhine-Westphalia
  - Universitätsklinikum des Saarlandes, Homburg/Saar, Saarland
  - AFL Arzneimittelforschung Leipzig GmbH, Leipzig, Sachen
  - ABX-CRO advanced pharmaceutical services Forschungsgesellschaft GmbH, Dresden, Saschen

REFERENCES:
- [Derived] Brashear HR, Ketter N, Bogert J, Di J, Salloway SP, Sperling R. Clinical Evaluation of Amyloid-Related Imaging Abnormalities in Bapineuzumab Phase III Studies. J Alzheimers Dis. 2018;66(4):1409-1424. doi: 10.3233/JAD-180675. PMID 30412493
- [Derived] Samtani MN, Xu SX, Russu A, Adedokun OJ, Lu M, Ito K, Corrigan B, Raje S, Brashear HR, Styren S, Hu C. Alzheimer's disease assessment scale-cognitive 11-item progression model in mild-to-moderate Alzheimer's disease trials of bapineuzumab. Alzheimers Dement (N Y). 2015 Oct 9;1(3):157-169. doi: 10.1016/j.trci.2015.09.001. eCollection 2015 Nov. PMID 29854935
- [Derived] Xu SX, Samtani MN, Russu A, Adedokun OJ, Lu M, Ito K, Corrigan B, Raje S, Brashear HR, Styren S, Hu C. Alzheimer's disease progression model using disability assessment for dementia scores from bapineuzumab trials. Alzheimers Dement (N Y). 2015 Jul 21;1(2):141-149. doi: 10.1016/j.trci.2015.06.005. eCollection 2015 Sep. PMID 29854934
- [Derived] Ketter N, Brashear HR, Bogert J, Di J, Miaux Y, Gass A, Purcell DD, Barkhof F, Arrighi HM. Central Review of Amyloid-Related Imaging Abnormalities in Two Phase III Clinical Trials of Bapineuzumab in Mild-To-Moderate Alzheimer's Disease Patients. J Alzheimers Dis. 2017;57(2):557-573. doi: 10.3233/JAD-160216. PMID 28269765
- [Derived] Liu E, Schmidt ME, Margolin R, Sperling R, Koeppe R, Mason NS, Klunk WE, Mathis CA, Salloway S, Fox NC, Hill DL, Les AS, Collins P, Gregg KM, Di J, Lu Y, Tudor IC, Wyman BT, Booth K, Broome S, Yuen E, Grundman M, Brashear HR; Bapineuzumab 301 and 302 Clinical Trial Investigators. Amyloid-beta 11C-PiB-PET imaging results from 2 randomized bapineuzumab phase 3 AD trials. Neurology. 2015 Aug 25;85(8):692-700. doi: 10.1212/WNL.0000000000001877. Epub 2015 Jul 24. PMID 26208959
- [Derived] Salloway S, Sperling R, Fox NC, Blennow K, Klunk W, Raskind M, Sabbagh M, Honig LS, Porsteinsson AP, Ferris S, Reichert M, Ketter N, Nejadnik B, Guenzler V, Miloslavsky M, Wang D, Lu Y, Lull J, Tudor IC, Liu E, Grundman M, Yuen E, Black R, Brashear HR; Bapineuzumab 301 and 302 Clinical Trial Investigators. Two phase 3 trials of bapineuzumab in mild-to-moderate Alzheimer's disease. N Engl J Med. 2014 Jan 23;370(4):322-33. doi: 10.1056/NEJMoa1304839. PMID 24450891